CLINICAL TRIAL: NCT01861223
Title: A Phase Ib Study of Afatinib Plus Nimotuzumab in Non-small Cell Lung Cancer Patients Who Progressed With Reversible EGFR TKI
Brief Title: Afatinib Plus Nimotuzumb for NSCLC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-11-087-007
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: NSCLC
Keywords: acquired resistance; gefitinib; erlotinib
MeSH Terms: interventions — Afatinib; nimotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- afatinib + nimotuzumab (Experimental)
  Interventions: Drug: afatinib (30 or 40mg) + nimotuzumab (100 or 200mg)

INTERVENTIONS:
Drug: afatinib (30 or 40mg) + nimotuzumab (100 or 200mg)

SUMMARY:
To find the optimal dose of afatinib and nimotuzumab in patients who acquired resistance to gefitinib or erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of stage IIIB or IV NSCLC
* Presence of EGFR sensitizing mutations (L858R mutation in exon 21 or exon 19 deletion) or response by RECIST on prior gefitinib or erlotinib or stable disease on prior gefitinib or erlotinib for at least 6 months
* Disease progression on treatemtn with gefitinib or erlotinib within 30 days
* Biopsy on disease progression
* Age ≥20 years
* ECOG performance status of 0, 1, or 2
* Measurable disease by the criteria of RECIST 1.1
* Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; creatinine clearance ≥ 45 mL/min

Exclusion Criteria:

* Known interstitial lung disease
* Prior treatment with EGFR targeting antibodies or BIBW 2992
* Prior three or more lines of chemotherapy for advanced NSCLC
* Significant bowel disease impairing drug absorption
* Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
* Have symptomatic, untreated, or uncontrolled central nervous system (CNS) metastases. Patients with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and corticosteroid use has been discontinued for at least 2 weeks prior to the first dose of study drug. Screening of asymptomatic patients without history of CNS metastases is not required.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose | 4 weeks
  To establish maximum tolerated dose (MTD) and recommended Phase II dose (RP2D) for BIBW 2992 and nimotuzumab in patients with acquired resistance to erlotinib or gefitinib

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea